CLINICAL TRIAL: NCT00328068
Title: Prospective, International, Multi-centre Study on ASAS Classification Criteria for SpA
Brief Title: Assessment of SpondyloArthritis Society (ASAS) Classification and Diagnostic Criteria for Early Axial Spondyloarthritis (SpA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, J. Sieper, Prof., Charite University, Berlin, Germany
Other Study IDs: ASAS-class-crit-1
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Spondyloarthritis; Spondylarthropathy; Spondylitis, Ankylosing
Keywords: ASAS classification; ASAS diagnostic criteria; spondyloarthritis; spondyloarthropathy; spondylitis, ankylosing; modified New York criteria for AS; ESSG criteria for SpA; Amor criteria for SpA; arthritis; enthesitis; magnetic resonance imaging
MeSH Terms: conditions — Spondylarthritis; Spondylarthropathies; Spondylitis, Ankylosing; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA will be collected in selected centres for analysis of candidate gene variants in ankylosing spondylitis/ spondyloarthritis. Serum and plasma sample will be collected for biomarker analysis with special focus on markers of bone metabolism
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Back pain / peripheral arthritis: Patients with chronic back pain of unknown origin and onset of back pain <45 years of age or patients with peripheral arthritis / enthesitis / dactylitis of unknown origin and onset <45 years of age

SUMMARY:
Background:

Existing criteria for AS/SpA such as mod. New York, ESSG, or Amor criteria for classification and/or diagnosis of spondyloarthritis have limitations when applied to early disease. Moreover, MRI is not part of any of the established criteria and the precise role of MRI in early axial disease has not been fully defined yet. Even less is known about sacroiliac (SI) changes in SpA patients with peripheral symptoms. A pilot study using data from 'paper patients' led to new candidate criteria for early spondyloarthritis. Subsequently, the members of the ASAS International Working Group decided to conduct a prospective multi-centre study to evaluate (validate) the new candidate criteria, and to assess their performance as diagnostic criteria.

Aims of the study:

1. To evaluate the new candidate criteria for axial SpA in a multi-centre setting.
2. To assess the potential role of the new candidate criteria to be used as diagnostic criteria. To accomplish this, inclusion of consecutive and undiagnosed patients is mandatory as are longer periods of follow-up .
3. To compare criteria encompassing the whole group of SpA such as ESSG and Amor criteria against criteria which are tailored to either predominant axial disease or predominant peripheral disease. To accomplish this, both patients with predominant axial disease (back pain) but also patient with predominant peripheral disease (arthritis/enthesitis) will be included.

DETAILED DESCRIPTION:
Background:

Existing criteria for AS/SpA such as mod. New York, ESSG, or Amor criteria for classification and/or diagnosis of spondyloarthritis have limitations when applied to early disease. Moreover, MRI is not part of any of the established criteria and the precise role of MRI in early axial disease has not been fully defined yet. Even less is known about sacroiliac (SI) changes in SpA patients with peripheral symptoms. A pilot study using data from 'paper patients' led to new candidate criteria for early spondyloarthritis. Subsequently, the members of the ASAS International Working Group decided to conduct a prospective multi-centre study to evaluate (validate) the new candidate criteria, and to assess their performance as diagnostic criteria.

Aims of the study:

1. To evaluate the new candidate criteria for axial SpA in a multi-centre setting.
2. To assess the potential role of the new candidate criteria to be used as diagnostic criteria. To accomplish this, inclusion of consecutive and undiagnosed patients is mandatory as are longer periods of follow-up .
3. To compare criteria encompassing the whole group of SpA such as ESSG and Amor criteria against criteria which are tailored to either predominant axial disease or predominant peripheral disease. To accomplish this, both patients with predominant axial disease (back pain) but also patient with predominant peripheral disease (arthritis/enthesitis) will be included.

Participating centres:

All ASAS members working in clinical practice are invited to participate in the study. More than one ASAS member/ rheumatologist per centre may participate.

Inclusion criteria:

Include newly referred patients if

* onset of symptoms (back pain / arthritis / enthesitis) < 45 years and
* undiagnosed* disease with the following symptoms:

  * chronic back pain (duration of back pain more than 3 months)
  * or / and peripheral arthritis (asymmetric arthritis / predominantly of the lower limbs)
  * or / and enthesitis
  * or / and dactylitis

    * Definition of 'undiagnosed':

The patient is being referred to your department because of chronic back pain, arthritis, enthesitis or dactylitis but has not been diagnosed confidently before by the referring physician/rheumatologist as having SpA or as definitely not having SpA. If the referring physician/GP/rheumatologist suspects SpA but is not certain about it, the patient is considered as undiagnosed.

Endpoints of the study:

* Primary endpoint: the diagnosis made by the rheumatologist (ASAS member) after the diagnostic work-up. This expert diagnosis serves as preliminary gold standard against which the various criteria will be compared. Final gold standard will be the outcome (diagnosis) after long-term follow up.
* Secondary endpoints: the diagnosis made by the rheumatologist at 2 and 5 years, respectively, after the first assessment. Thus, all patients should be invited to follow-up visits after 2 and 5 years, respectively.

Further study rules:

* Include all newly referred patients strictly consecutively as long as they meet the inclusion criteria.
* The decision to include a patient should be based solely on the fulfilment of the inclusion criteria, and should be made ideally before you make the final diagnosis (prospective study design).
* Patients who have been diagnosed confidently and correctly by the referring physician prior to being referred to your department cannot be included in the study.
* If you are unable to perform MRIs in your clinical setting you cannot include patients with undiagnosed chronic back pain.
* If you want to include patients with undiagnosed chronic back pain, perform MRI of sacroiliac (SI) joints in the first 10 patients with axial SpA and in the first 10 patients with non-SpA related (mechanical) back pain. In subsequent patients you may perform MRIs as needed on clinical grounds. (Explanation: a minimum number of MRIs in both SpA and non-SpA patients from several centres is necessary to obtain reliable results on sensitivity and specificity of MRI in early axial SpA.)
* MRI of SI joints in patients with peripheral symptoms only will be performed in selected centres (centres already indicated whether this will be possible).
* MRI results will be taken as provided by the local centre (either read by the radiologist or rheumatologist, whoever has greater experience). Results will be categorized into 'presence or absence of active inflammatory lesions compatible with SpA', and 'presence or absence of chronic lesions compatible with sacroiliitis/spondylitis'. (Selected centres will be invited to send us their MRIs for validation of locally performed readings (the intention is to increase the quality of data).
* Plain radiographs of the SI joints and lumbar spine are mandatory in all patients with undiagnosed chronic back pain. Previously taken radiographs are acceptable if they are not older than 6 months. Results are taken as provided locally either by the radiologist or rheumatologist, whoever has greater experience.
* At the end of the diagnostic work up, a preliminary diagnosis must be made by the ASAS rheumatologist as is done in usual daily clinics. It is not important to be absolutely confident about the diagnosis at this stage since this i) reflects daily practice, and ii) the level of confidence with the diagnosis will be assessed as well. (It is more important to include all patients consecutively in your centre in order to avoid any selection bias.) The senior ASAS member should supervise other physicians experienced in SpA in her/his department who participate in the study.
* Patients with peripheral symptoms should be included if they meet the inclusion criteria. Patients with peripheral symptoms and a history of chronic back pain or with concomitant chronic back pain must undergo radiographic examination of the SI joints. Patients with non-specific musculoskeletal pain or arthralgia (without arthritis) only cannot be included.

Data documentation:

The results of the clinical history, physical examination, blood tests, radiographs, and MRIs, and the diagnosis will be entered into the CRF locally by the ASAS member during/after the diagnostic work-up. The diagnosis will be made by the local rheumatologist (ASAS member or an experienced colleague at the centre). The completed CRF should be sent to the coordinating centre (Berlin) for data check and data entry. A copy of the CRF should remain locally at the study centre. The name, date of birth, address, and telephone number must also be kept locally in the centre since follow-up assessments after 2 years and after 5 years are planned.

Sample size and inclusion period:

It is estimated that about 400-500 patients with SpA (ca 250-300 axial and 150-200 peripheral SpA) with complete data sets are needed to allow for a reliable comparison of new candidate criteria with established criteria. Since the prevalence of SpA among newly referred patients with unclear diagnoses varies from centre to centre any calculation of the control group size (and thus total sample size) is bound to be inaccurate. Therefore, the proposal is that each centre recruits as many consecutive patients as possible until indicated by the study coordinators to stop inclusion. The study coordinators can adequately terminate the inclusion period only if the completed CRFs are sent within a reasonably short period of time (< 2 weeks) to the coordinating centre. Data entry and data analysis will be done at the coordinating centre.

DNA/RNA-analysis and biomarker analysis:

In addition to the clinical study which aims to arrive at new classification and diagnostic criteria, two groups of researches will perform laboratory experiments in patients from selected centres: Genetic polymorphisms and gene products (RNA) which are potentially associated with spondyloarthritis will be analysed by Prof. Matthew Brown in Brisbane, Australia. A second group of researchers (Prof. Walter Maksymowych, Canada, Prof. Mikkel Ostergaard, Denmark, Prof. Rob Inman, US, and Prof. David Yu, US) will analyse several biomarkers such as cartilage break-down or bone formation proteins in serum and/or plasma. Data from both experimental projects may be of potential diagnostic value in the future and/or may reveal novel insights into pathophysiological mechanisms of spondyloarthritis.

Longterm follow-up:

A second follow-up visit of all patients 2 years after the first encounter and also 5 years after the first encounter is highly warranted since diagnoses may change over time and the final diagnosis after long-term follow up is the most important gold standard. Thus, a record containing the names, addresses, and phone numbers of all patients included in the study must be stored locally at the study site. The patient is best informed at the first visit that a follow-up assessments 2 and 5 years later are envisaged.

ELIGIBILITY:
Inclusion Criteria:

Include newly referred patients if:

* Onset of symptoms (back pain/arthritis/enthesitis) < 45 years
* Undiagnosed disease with the following symptoms:

  * chronic back pain (duration of back pain more than 3 months)
  * and/or peripheral arthritis (asymmetric arthritis/predominantly of the lower limbs)
  * and/or enthesitis
  * and/or dactylitis

Exclusion Criteria:

* No symptoms such as specified in inclusion criteria: back pain, arthritis, enthesitis
* Definite diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic back pain of unknown origin or peripheral arthritis / enthesitis / dactylitis of unknown origin who are referred to a rheumatologist for diagnostic work-up
Sampling Method: Non-Probability Sample
Enrollment: 992 (Estimated)
Dates: Start 2006-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Spondyloarthritis | 2 years

SECONDARY OUTCOMES:
Patients with a retained diagnosis of spondyloarthritis after follow-up | 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rudwaleit, MD, Principal Investigator — Universitatsmedizin Berlin, Charité Campus Benjamin-Franklin, Med. Clinic I, Rheumatology, Hindenburgdamm 30, 12200 Berlin, Germany; Joachim Sieper, MD, Principal Investigator — Charité Universtaetsmedizin Berlin
Locations (35):
- Case Western Reserve University at MetroHealth Medical Centre, Cleveland, Ohio, United States
- University Hospital Gent, Ghent, Belgium
- Rheumatology Division, São Paulo, Brazil
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - The Toronto Hospital, Toronto, Ontario
- China (2):
  - Chinese PLA General Hospital, Beijing
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
- Division of Rheumatology, Bogotá, Colombia
- Hvidovre Hospital, University of Copenhagen, Hvidovre, Denmark
- France (2):
  - Service de Rheumatologie, Marseille
  - Rheumatology B Department, Paris
- Germany (3):
  - Brandt, Berlin
  - Universitaetsmedizin Berlin, Charité Campus Benjamin-Franklin, Med. Clinic I, Rheumatology, Hindenburgdamm 30, Berlin
  - Rheumazentrum Ruhrgebiet, Herne
- Géher, Budapest, Hungary
- Seroja Rheumatic Centre, Semarang, Indonesia
- St. Vincent's Hospital, Dublin, Ireland
- Italy (3):
  - University of Florence, Florence
  - Arcispedale S. Maria Nouva, Reggio Emilia
  - Caterina Naclerio, Scafati (SA)
- Hospital General de México, Mexico City, Mexico
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Kennemer Gasthuis, Locatie Deo, HG IJmuiden
  - University Hospital Maastricht, Maastricht
- Spain (2):
  - Hospital Universitario "Reina Sofia", Córdoba
  - Hospital Universitario Gregorio Marañón, Madrid
- Balgrist University Hospital, Zurich, Switzerland
- Taiwan (2):
  - Veterans General Hospital Taipei, Beitou Dist. Taipei
  - Wei, Taichung
- Turkey (Türkiye) (3):
  - Duruöz, Bornova
  - Division of Rheumatology, Elâzığ
  - Izmir University Hospital, Izmir
- United Kingdom (3):
  - Glasgow Royal Infirmary, Queen Elizabeth Building, Glasgow
  - King George Hospital, Goodmayes
  - ChapelChapel Allerton Hospital, Leeds

REFERENCES:
- [Background] Rudwaleit M, Metter A, Listing J, Sieper J, Braun J. Inflammatory back pain in ankylosing spondylitis: a reassessment of the clinical history for application as classification and diagnostic criteria. Arthritis Rheum. 2006 Feb;54(2):569-78. doi: 10.1002/art.21619. PMID 16447233
- [Background] Rudwaleit M, Sieper J. Positive and negative predictive values from published studies can be misleading for decision-making in clinical practice. Rheumatology (Oxford). 2006 Jun;45(6):779-80; author reply 780-1. doi: 10.1093/rheumatology/kel083. Epub 2006 Apr 4. No abstract available. PMID 16595519
- [Derived] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- See also: ASAS is an international society of experts in the field of spondyloarthritis. — http://www.asas-group.org/